CLINICAL TRIAL: NCT00533754
Title: Y402H Comlement Factor H Polymorphism and Age-Related Macular Degeneration in the Austrian Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rudolf Foundation Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: EK 06-076-VK; EK 06-076-VK
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2007-09-21 (Estimated); Status verified 2007-09

CONDITIONS: Age-Related Macular Degeneration
Keywords: age-related macular degeneration, genetics
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: drawing blood

SUMMARY:
The aim of the study is to show a higher expression of the Y402H polymorphism in the complement factor H in patients with AMD compared to healthy individuals.

Additionaly a correlation between a subsided infection with chlamydia and patients with AMD and a factor H polymorphism will be investigated. An interrelationship with the VEGF-plasma level shall give more hints into the pathomechanism of AMD.

ELIGIBILITY:
Inclusion Criteria:

* man and women over 18 years old
* Filled out informed consentBereitschaft zur Teilnahme
* Diagnosis of non-exudative/ exudative age related macular dgeneneration

Exclusion Criteria:

* inherited retinal diseases
* other aquired retinal/ macular
* missing informed consent

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-07; Study Completion 2007-11 (Estimated)

PRIMARY OUTCOMES:
higher expression of the Y402H polymorphism in the complement factor H in patients with AMD compared to healthy individuals

SECONDARY OUTCOMES:
a correlation between a subsided infection with chlamydia and patients with AMD and a factor H polymorphism will be investigated. An interrelationship with the VEGF-plasma level shall give more hints into the pathomechanism of AMD

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Binder, M.D., Study Chair — Rudoulf Foundation Clinic
Locations (1):
- Rudoulf foundation Clinic, Vienna, Vienna, Austria